CLINICAL TRIAL: NCT07100743
Title: A Randomised Double-blind Placebo-Controlled Trial of Multi-Strain Probiotic Supplementation (Hexbio®) in Malaysian Patients With Drug-Resistant Epilepsy (ProbE)
Brief Title: Trial of Multi-Strain Probiotic Supplementation (Hexbio®) in Malaysian Patients With Drug-Resistant Epilepsy (ProbE)
Acronym: ProbE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: B-Crobes Laboratory Sdn. Bhd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: JEP-2023-151; FF- 2023-132 (Other Grant/Funding Number: National University of Malaysia); FF- 2023-132 (Other Grant/Funding Number: B-Crobes Laboratory Sdn Bhd)
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Epilepsies Refractory
Keywords: drug-resistant epilepsy, quality of life, seizure worry, emotional well-being, probiotic, Malaysia
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: The participants are randomized to receive either HEXBIO MCP Granule probiotic or placebo. Patients will be instructed to consume one sachet directly before meal (drink water if needed) twice daily, for two months. The placebo sachets will contain the same ingredient as the probiotic sachet but without the Lactobacillus sp. and Bifidobacterium sp. Participants in the placebo group will receive an identical Hexbio sachet (aluminum foil sachet.) with non-microbial material.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): HEXBIO MCP Granule probiotic is prepared in sachets which consist of the following probiotics: Lactobacillus acidophilus (BCMC 1 12130)107mg, Lactobacillus casei (BCMC 1 12313) -107mg, Lactobacillus lactis (BCMC 1 12451)-107 mg, (BCMC 1 02290) -107mg, Bifidobacterium infantis (BCMC 1 02129) -107mg and Bifidobacterium longum (BCMC 102120)-107mg. Patients will be instructed to consume one sachet directly before meal (drink water if needed) twice daily, for two months.
  Interventions: Dietary Supplement: Probiotic Agent
- Placebo (Placebo Comparator): The placebo sachets will contain the same ingredient as the probiotic sachet but without the Lactobacillus sp. and Bifidobacterium sp. Participants in the placebo group will receive an identical Hexbio sachet (aluminum foil sachet.) with non-microbial material.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Agent — HEXBIO MCP Granule probiotic is prepared in sachets which consist of the following probiotics: Lactobacillus acidophilus (BCMC 1 12130)107mg, Lactobacillus casei (BCMC 1 12313) -107mg, Lactobacillus lactis (BCMC 1 12451)-107 mg, (BCMC 1 02290) -107mg, Bifidobacterium infantis (BCMC 1 02129) -107mg and Bifidobacterium longum (BCMC 102120)-107mg
  Other Names: Hexbio
  Arms: Intervention
Dietary Supplement: Placebo — The placebo sachets will contain the same ingredient as the probiotic sachet but without the Lactobacillus sp. and Bifidobacterium sp. Participants in the placebo group will receive an identical Hexbio sachet (aluminum foil sachet.) with non-microbial material.
  Arms: Placebo

SUMMARY:
Probiotics are good, live bacteria and/or yeast, that live in our guts and causes no harm. They help in digestion and overall well-being of our gut system. The purpose of the study is to assess the effect of probiotics on the quality of life and seizure frequency in epilepsy patients with uncontrolled seizures.

This experimental study involves an interview by the researchers from UKM for the demographic of epilepsy, seizure control and quality of life using a questionnaire. The questionnaire will take about 15 minutes to complete, and you will need to answer all questions without assistance.

You will be randomized either into the active group or the placebo group. If you are in the active group, you will need to take one HEXBIO MCP Granule probiotics sachet directly before meal (drink water if needed) twice daily, for two months, in addition to your pre-existing epilepsy treatment. The HEXBIO MCP Granule probiotic consists of the following probiotics: Lactobacillus acidophilus, Lactobacillus casei, Lactobacillus lactis, Bifidobacterium infantis and Bifidobacterium longum. Initially, some people may experience temporary mild gastrointestinal symptoms such as abdominal cramping, soft stools and flatulence as body adapts to the introduction of friendly bacteria. The symptoms will subside gradually after few days.

If you are in the placebo group, you will also need to take one sachet twice daily before meal, for two months, in addition to the epilepsy treatment. The placebo sachets will contain the same ingredient as the probiotic sachet but without the Lactobacillus sp. and Bifidobacterium sp. The placebo sachet is also to be taken the same way as the probiotic sachet.

At two months of follow up, you will be interviewed once again to assess the changes of seizure frequency (using seizure diary), quality of life and the adverse effects of experienced. A sachet-count (using sachet diary) will also be done to assess the compliance.

Benefits This study is done in an attempt to assess the changes in quality of life and seizure frequency in patients with refractory epilepsy as compared to the control group.

Risks There is no risk in this study. All information disclosed during this study is strictly confidential. You do not have to pay to participate in this study.

If seizure or quality of life worsened during this period, you will be referred to the respective team for the optimization of anti-seizure medications.

Do you have to take part? Participation in this study is voluntary. If you agree to take part, then you will be asked to sign the "informed Consent Form". Should you decide to participate, you can still withdraw at any time during the study without penalty. Your data will be discarded and not be used. Regardless of your decision at any point in time, your treatment will not be affected.

Data and Confidentiality The data in this study will be made into a report which may be published. The data will be reported in a collective manner with no reference to an individual. Hence your identity will be kept confidential. There is no conflict of interest among the researchers.

DETAILED DESCRIPTION:
Epilepsy is a chronic neurological disorder, characterized by two or more unprovoked seizures occurring more than 24 hours apart owing to excessive or asynchronous brain neuronal activities. It has a high global prevalence whereby the overall lifetime prevalence is 7.6 per 1,000 populations worldwide.1 Similarly, in Malaysia, the prevalence of epilepsy is up to 7.8 in 1,000 populations. 2

The mainstay of treatment for all types of epilepsy is anti-seizure medications (ASM). There are many types of ASM that are being used currently, ranging from a narrow to a broad spectrum. In spite of this, only 70% of patients on single ASM are able to achieve seizure-free. The remaining one third will need an addition or substitution of ASM.2

Refractory epilepsy is defined as persistent seizures despite being on optimal dose of two or more ASM. The standard treatment for refractory epilepsy includes ASM polytherapy and non -pharmacological methods. The choice of ASM includes medications such as phenytoin, valproate, carbamazepine, topiramate, levetiracetam, lacosamide, lamotrigine, oxcarbazepine, clonazepam, eslicarbazepine, zonisamide and perampanel. Ketogenic diet, surgery, and neurostimulator implantation were the non-pharmacological alternatives employed on these patients but only showed minimal effectiveness.3 If left untreated, it is associated with a poor quality of life (QoL), higher mortality rate, and increased socio-economic burden.

In recent years, the interest in probiotics was at all-time high in Western countries and China. The bidirectional relationship between the gut microbiota and brain, also known as the 'microbiota-gut-brain axis' has gained the attention of many, especially in those related to Parkinson's disease, autism spectrum disorders (ASD), schizophrenia, and multiple sclerosis. Probiotics improved non-motor symptoms in Parkinson's Disease. 4Probiotics as an adjunctive were also proven to prevent the somatic symptoms in schizophrenia and improve autistic symptoms in autism spectrum disorder. 5-7

Probiotics had been used in preclinical and clinical research contexts and shown positive effects on early life stress-induced anxiety and depression-related behavior in rodents, however specific mechanism remains unknown.8,9The 'microbiota-gut-brain axis' is a complex interaction involving the neuroendocrine, immunological and direct neural mechanisms. It is hypothesized that microbes and their metabolites alter the transport of neuroactive chemicals into the nervous system thus increasing the permeability of the gut wall and allowing the psychoactive chemicals to enter the blood and subsequently to the brain. 10-13

The use of probiotics in improving the quality of life of patients with refractory epilepsy have also been explored recently. Gomez et.al., proved that the use of probiotics caused a reduction in seizure frequency in more than a quarter of patients with refractory epilepsy leading to an improved quality of life. 11 Likewise, Wang et.al., demonstrated that probiotics improved seizure control, anxiety and depression in temporal lobe epilepsy, thus a better quality of life.14

Probiotics are defined as live microorganisms that confers a health benefit to the host when administered in the adequate amount. 10 The commonly seen probiotics are grouped into Lactobacillus, Bifidobacterium and Saccharomyces, which are seen in our human gut. Probiotics have been safely used in many studies. Only a minority have suffered from mild gastrointestinal symptoms, namely abdominal cramping, nausea, soft stools, flatulence and taste disturbances. 15

To our best knowledge, there are still limited papers with regards to probiotics and epilepsy, especially in our Malaysian setting. Hence, by conducting this study, to study the effects of probiotics as an adjunctive treatment in patients with refractory epilepsy. We hope that the findings from this study could shed some light on the treatment for refractory epilepsy in our setting.

CHAPTER 2.0 - PROBLEM STATEMENT & OBJECTIVES Problem Statement

1. Does quality of life improve post administration of probiotics in refractory epilepsy patients compared to the placebo group?
2. Does a lower occurrence of seizure seen post administration of probiotics in refractory epilepsy patients compared to the placebo group?

Primary Objective

1. To compare the quality of life score pre- and post-administration of probiotics inter- and intragroup of refractory epilepsy patients.

Secondary Objective 1. To assess the frequency of seizure pre- and post- administration of probiotics inter- and intragroup of refractory epilepsy patients.

Hypotheses

1. The quality of life score improves post administration of probiotics in refractory epilepsy patients compared to the placebo group.
2. There is a reduction in the seizure frequency post administration of probiotics in refractory epilepsy patients compared to the placebo group.

CHAPTER 3.0 - METHODOLOGY 3.1 Study Design This is a single center, double blinded, placebo controlled, case controlled clinical trial.

3.2 Sample Size The sample size for this study is calculated using the sample size for two mean quantitative data by Rosner, B., from Fundamentals of Biostatics. 16

N = (Zα/2 +Zβ)2 δ2 d2 in which, N : Number of samples required Zα/2 : probability of falsely rejecting a true null hypothesis (). The critical value of the normal distribution at α/2 (for a confidence level of 95%, α is 0.05 and the critical value is 1.96) Zβ : probability of failing to reject a false null hypothesis (β). The critical value of the normal distribution at β (for a power of 80%, β is 0.2 and the critical value is 0.84) δ : Standard deviation obtained from previous study or pilot study d : an average difference between the intervention and control group (d = u1 - u2/2)

Using a recent study finding, 14 Seizure reduction of 1-30% (probiotics vs. placebo: 31.4% vs. 5.7%, p < 0.05) with mean difference of 25.7 and the standard deviation of the two groups is estimated 20%.

The QOLIE-89 scores had standard deviation of probiotics vs. placebo: 60.29 ± 14.01 vs. 51.91 ± 13.20, p = 0.006) with mean difference of 8.38 and standard deviation of 14.

The minimum sample size needed for each group to detect whether the stated difference exists between the two means (with the required confidence level and power) is 44, for seizure reduction.

Whereas, the minimum sample size needed for each group to detect whether the stated difference exists between the two means (with the required confidence level and power) is 10, for Quality of Life.

3.3 Inclusion and Exclusion Criteria(s)

*The inclusion and exclusion criteria for both the probiotic and control groups are similar.

Inclusion Criteria(s)

1. Patients diagnosed with refractory focal epilepsy
2. Have at least one self-reported seizure per month
3. On two or more ASM
4. Aged 18 years and above, who is able to read and write in English and/or Bahasa Malaysia
5. Provide informed consent

Exclusion Criteria

1. Had status epilepticus in the last 12 months
2. Changes in ASM dose or type in the 30 days prior to inclusion to this study
3. Seizures related to alcohol / drug abuse / metabolic cause / infections.
4. Use of probiotics, immune-suppressants, prolonged antibiotics (more than 2 weeks), traditional treatment, supplements in the 30 days before the inclusion of the study.
5. Gastrointestinal related diseases such as lactose intolerance, coeliac disease
6. Renal or hepatic insufficiency (Based on recent six-month blood profile)
7. Progressive neurological disease (Alzheimer's disease, Parkinson's Disease, Motor Neuron Disease)
8. Pregnancy

3.4 Study Population Patients diagnosed with refractory epilepsy attending the Neurology Clinic in Hospital Canselor Tuanku Mukhriz (HCTM), Cheras, Kuala Lumpur.

3.5 Recruitment/Data Collection The study will be conducted in HCTM Neurology Clinic starting from 3rd April 2023 till 2 March 2026.

For this study, patients will be selected based on the inclusion criteria(s). We will randomize the patient selection to avoid confounding between treatment effects and other unknown effects. The eligible patient will be assigned to group A (Active) and the next patient recruited will be assigned to the group B (Placebo) until 57 patients in each arm is met. The subjects are followed and outcomes are recorded. Both researcher and sample recruited are blinded (double-blind clinical trial with random selection of patients. Informed consent will be obtained from the patient. They will be interviewed using the designated questionnaire. The questionnaire consists of social demographic data, past medical history, characteristics of epilepsy, seizure frequency and types of ASM, which are taken at baseline.

Patients will be randomized to either the active group or placebo group. For the active group, patients will be given HEXBIO MCP Granule probiotics one sachet twice daily for two months. As for the placebo group, the patients will be given placebo, also to be taken one sachet twice daily for two months. There is no difference between the treatment or placebo sachet appearance (color, size). Both groups will be instructed to continue their current epilepsy treatment.

At baseline, the patients from both groups will be assessed for seizure frequency using a seizure diary, type of ASM, and quality of life questionnaire. The Quality of Life will be assessed using the questionnaire quality of life in epilepsy-31 (QOLIE-31), both in English and Malay. On review after two months, the patients from both groups will be assessed for changes in seizure frequencies (using seizure diary) and adherence to ASM, and Quality of Life. Adherence to intervention (probiotics/placebo) will also be assessed via sachet count (using sachet diary) at the end of two months. Patients who missed probiotics or placebo for 14 days and more will be dropped out from the study. In case of worsening seizure frequency, the anti-seizure medications will be adjusted accordingly as per usual seizure management protocol.

3.6 Study Tools Questionnaire For the purpose of this study, we will be using the self-administered, validated quality of life in epilepsy questionnaire (QOLIE-31), which comprises of 7 components: energy, emotional well-being, daily activities, mental activity, medication effects, worry and overall quality of life. QOLIE-31 was designed to evaluate the QoL of all patients with epilepsy. This screening tool have been widely used in many studies. Patients will be given an option to choose either the English or Malay version of the questionnaire based on their language proficiency. Both the epilepsy questionnaires have been validated and permission obtained. (Appendix D and E)

The scoring system for each item range from 0-6, and the overall score will be calculated based on weighting and summing QOLIE-31 scale scores as per the formula mentioned in the scoring sheet. The higher the score, the better the quality of life.

Intervention HEXBIO MCP Granule probiotic is prepared in sachets which consist of the following probiotics: Lactobacillus acidophilus (BCMC 1 12130)107mg, Lactobacillus casei (BCMC 1 12313) -107mg, Lactobacillus lactis (BCMC 1 12451)-107 mg, (BCMC 1 02290) -107mg, Bifidobacterium infantis (BCMC 1 02129) -107mg and Bifidobacterium longum (BCMC 102120)-107mg. Patients will be instructed to consume one sachet directly before meal (drink water if needed) twice daily, for two months. There are no known contraindications reported. According to the Monthly Index of Medical Specialties (MIMS), there are no drug -drug interactions with ASM except that when taken with antibiotics. Similarly, there are no documented interactions between probiotics and phenobarbitone. 17 During the study, patients need to avoid taking any health supplements except HEXBIO. If they are required to take antibiotics at any time point of the study, they should inform the respective investigator.

The placebo sachets will contain the same ingredient as the probiotic sachet but without the Lactobacillus sp. and Bifidobacterium sp. Participants in the placebo group will receive an identical Hexbio sachet (aluminum foil sachet.) with non-microbial material. The placebo sachet is also to be taken the same way as the probiotic sachet. Both group of patients (active and placebo) will be given the exact number of sachet and seizure diary and upon two months of assessments, they are required to bring back all used sachets and seizure diary for documentation purpose.

3.7 Data Analysis All the data collected will be kept in a patient data collection sheet and analysis will be conducted using Statistical Product and Service Solution (SPSS) version 26. Descriptive statistics will be used to present background and study variables.

Analysis will be done using intention-to-treat (ITT). After recording analysis of 50% of the patients, if a positive changes in seizure reduction and quality of life are seen, an interim analysis will be done. The probiotics effectiveness is described as more than 50% reduction in seizures during the treatment as compared to baseline. Kolmogorov-Smirnov test will be conducted to assess the normality of the data. Then bivariate (t-test/Mann Whitney U test/compare paired t-test) and multivariate analysis (Multiple Linear Regression) will be conducted. The association will be considered significant if the p value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria(s)

  1. Patients diagnosed with refractory focal epilepsy
  2. Have at least one self-reported seizure per month
  3. On two or more ASM
  4. Aged 18 years and above, who is able to read and write in English and/or Bahasa Malaysia
  5. Provide informed consent

     Exclusion Criteria

  <!-- -->

  1. Had status epilepticus in the last 12 months
  2. Changes in ASM dose or type in the 30 days prior to inclusion to this study
  3. Seizures related to alcohol / drug abuse / metabolic cause / infections.
  4. Use of probiotics, immune-suppressants, prolonged antibiotics (more than 2 weeks), traditional treatment, supplements in the 30 days before the inclusion of the study.
  5. Gastrointestinal related diseases such as lactose intolerance, coeliac disease
  6. Renal or hepatic insufficiency (Based on recent six-month blood profile)
  7. Progressive neurological disease (Alzheimer's disease, Parkinson's Disease, Motor Neuron Disease)
  8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | 2 months
  To compare the quality of life score pre- and post-administration of probiotics inter- and intragroup of refractory epilepsy patients

SECONDARY OUTCOMES:
Seizure Frequency | 2 months
  To assess the frequency of seizure pre- and post- administration of probiotics inter- and intragroup of refractory epilepsy patients

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the journal requirements